CLINICAL TRIAL: NCT00942240
Title: A Phase I, Double-Masked, Multiple Rising Dose Study of ACU-4429 in Healthy Male and Female Subjects
Brief Title: Safety and Tolerability of Repeat Doses of ACU-4429 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8211 725
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
MeSH Terms: interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACU-4429 tablet (Experimental)
  Interventions: Drug: ACU-4429
- matching placebo tablet (Placebo Comparator)
  Interventions: Drug: matching placebo tablet

INTERVENTIONS:
Drug: ACU-4429 — administered orally once a day for 14 days
  Arms: ACU-4429 tablet
Drug: matching placebo tablet — administered orally once a day for 14 days
  Arms: matching placebo tablet

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of repeated doses of a new investigational drug (ACU-4429) in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* males or females, between 25 and 55 years of age, inclusive
* within BMI range 19 to 32 kg/m2 at Screening
* in good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs;
* clinical laboratory evaluations (including serum for Chem-20 [fasted at least 10 hours], CBC with differential and platelet counts, PT, INR, and aPTT, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator;
* Males (or female partners of male subjects)and females must be sterile, or agree to use approved contraceptive measures throughout the study period and 45 days after the End of In House Study.
* able to comprehend and willing to sign an Informed Consent Form.

Exclusion Criteria:

* significant history or clinical manifestation of any significant metabolic, endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator);
* history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
* history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs, except that appendectomy, hernia repair, and/or cholecystectomy will be allowed;
* history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant;
* participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to Check-in;
* Is currently using, or has recently received treatment with a medication disallowed by the Protocol.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse events, physical exam, ECG, vital signs, laboratory tests and visual tests | 20 days

SECONDARY OUTCOMES:
Pharmacokinetics as measured by plasma ACU-4429 drug levels | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: William Lewis, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States